CLINICAL TRIAL: NCT04878640
Title: Sleeve Gastrectomy and Cholecystectomy Are Safe in Obese Patients With Asymptomatic Cholelithiasis: A Multicenter Randomized Trial
Brief Title: Sleeve Gastrectomy and Cholecystectomy Are Safe in Obese Patients With Asymptomatic Cholelithiasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer Alsaied Alnaimy, assistant professour of general and laparoscopic surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sleeve Gastrectomy
Record Dates: First submitted 2021-05-01; First posted 2021-05-07 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Bariatric Surgery Candidate
Keywords: obesity; bariatric surgery; concomitant, cholecystectomy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): patients with morbid obesity and gall bladder stone underwent concomitant laparoscopic cholecystectomy in the same setting during laparoscopic sleeve gastrectomy
  Interventions: Procedure: patients with morbid obesity and gall bladder stone underwent concomitant laparoscopic cholecystectomy in the same setting during laparoscopic sleeve gastrectomy
- Group B (Active Comparator): patients with morbid obesity and gall bladder stone underwent laparoscopic sleeve gastrectomy without concomitant laparoscopic cholecystectomy
  Interventions: Procedure: patients with morbid obesity and gall bladder stone underwent laparoscopic sleeve gastrectomy without concomitant laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: patients with morbid obesity and gall bladder stone underwent concomitant laparoscopic cholecystectomy in the same setting during laparoscopic sleeve gastrectomy — patients with morbid obesity and gall bladder stone underwent concomitant laparoscopic cholecystectomy in the same setting during laparoscopic sleeve gastrectomy
  Arms: Group A
Procedure: patients with morbid obesity and gall bladder stone underwent laparoscopic sleeve gastrectomy without concomitant laparoscopic cholecystectomy — patients with morbid obesity and gall bladder stone underwent laparoscopic sleeve gastrectomy without concomitant laparoscopic cholecystectomy
  Arms: Group B

SUMMARY:
Introduction:

Obesity is an increasingly serious public health problem on a global level. Gallstones may become symptomatic after sleeve gastrectomy surgery. There is a debate regarding concomitant cholecystectomy during bariatric surgery.

Aim of the study: This study analyzed outcomes of laparoscopic sleeve gastrectomy (LSG) with and without concomitant laparoscopic cholecystectomy in morbid obese patients with gall bladder stones.

Patients and methods: We conducted randomized clinical study on 222 patients. These patients were categorized into two equal groups (111 in each group) .Group A: underwent SG and concomitant laparoscopic cholecystectomy in morbid obese patient with evidence of gall bladder stone, Group B: SG only without concomitant LC inspite of evidence of gall bladder stone. This study was performed at single institution from January 1, 2016 to January 1, 2019.

DETAILED DESCRIPTION:
The WHO (World Health Organization) has already affirmed that obesity is a universal epidemic that represents one of the substantial present health complications . Bariatric surgery (BS) is the pillar of cure for morbid obesity with thousands of surgeries implemented each year .Bariatric surgery guides patients to waste weight and correct obesity- related troubles, and improves quality of life .Sleeve Gastrectomy (SG) materialized as the first part of a staged duodenal switch step and afterwards changed to be a main restrictive bariatric surgery .The comprehensive pervasiveness of cholelithiasis in the normal populace is 10% to 20%. The pervasiveness of cholelithiasis in patients with severe obesity is 3 to 5 times greater in comparison with that for gangly persons .In obese patients, gallstone is more emlematic than in non-obese people .

Aim of the work, gap statement and strength of the study:

During laparoscopic sleeve gastrectomy for morbid obesity surgery, there is no golden standard of dealing with gall bladder stones, which is generally selected by the surgeon's preferences or by local conditions. For many surgeons, the benefit of routine cholecystectomy in patients with gall bladder stones did not justify an additional risk and the risks of cholecystectomy after a laparoscopic sleeve gastrectomy may be higher due to adhesion and expose patients to another surgery. Others believe that concomitant cholecystectomy may increase operative time, morbidity and decrease fat after laparoscopic sleeve gastrectomy helps good identification of anatomy during later laparoscopic cholecystectomy. In this study, we have designed a randomized clinical trial to compare outcomes in patients who underwent laparoscopic sleeve gastrectomy with or without concomitant laparoscopic cholecystectomy in patients with gall bladder stones (Symptomatic or asymptomatic). The primary aim was to compare the morbidity and mortality rate during and after both techniques. The secondary aim was to evaluate the postoperative body weight. The tertiary aim was to detect the incidence of symptomatic and asymptomatic gall bladder stone in cases with no concomitant laparoscopic cholecystectomy.

2. Material and methods

Study design:

A prospective randomized controlled clinical study was conducted in bariatric surgical unit of our University Hospital (single center) between January 2016 to January 2019. Patients were admitted with clinical diagnosis of morbid obesity with gall bladder stone. A total of 222 patients were randomly divided into two groups: Group A (n=111), patients with morbid obesity and gall bladder stone underwent concomitant laparoscopic cholecystectomy in the same setting during laparoscopic sleeve gastrectomy. Group B (n=111), patients with morbid obesity and gall bladder stone underwent laparoscopic sleeve gastrectomy without concomitant laparoscopic cholecystectomy. it is a simple random sample with a balance. Sample size was calculated to be 222 (111 in each group) according to the following data: the morbidity in Group A (LSG+CC) was 18.75% compared to 6.25% in Group B (LSG) at confidence level 95%, power 80% using Open.Epi. The selection of patients was done by simple random technique. Each included patient was taken number from one to 222 and randomization was done using random table where odds numbers for Group A and even numbers for Group B to avoid bias in the this study.

Method of randomization: Patients were randomly allocated using a random sequence generator. Random allocations were sequentially numbered in sealed opaque envelopes, which were opened during surgery before carrying out the surgery. Patients were undiscerning to the assigned group until the study was completed. It is done by recording service.

The work has been reported in line with consolidated standards of reporting trials (CONSORT) guidelines .

Patient selection criteria:

To be eligible for the study, patients had to fulfill all the consecutive principles: Male and Non pregnant female, >20 years old, All patients were contender for bariatric surgery in conformity with National Institutes of Health consensus criteria for the management of morbid obesity (BMI ≥ 40 kg/m² or BMI ≥ 35 kg/m² with compelling co-morbidities linked to obesity),, had pre-operative ultrasound and patients who completed at least two-years follow up. Omission criteria were younger than 20 years, History of cholecystectomy, No pre-operative imaging available within 6 months, dearth of interest. Subjective mess and cognitive vulnerability that halt the patient from considering the operation, Drug or alcohol junkie, Patients unsuitable for general anesthesia, preceding bariatric operation, Patients with calcular obstructive jaundice underwent ERCP with stenting and Cases with arduous displaying of right upper quadrant or liver cirrhosis found at surgery.

Types of outcome and measurement (study endpoints):

Primary outcomes were the total postoperative morbidities and mortality(within 30 days and 90 days postoperative): including time of operation (in minutes), intraoperative blood waste (ml), Vascular/visceral damage at operation, Hematoma/Seroma , Length of hospital stay (in days) , Wound infection at any time point , rehabilitation time to normal activity (in days), In-hospital mortality , ICU/days (intensive care unit admission) and hospital length of stay (days) , postoperative ileus and postoperative stricture. Secondary outcomes were postoperative BMI, percent excess BMI loss (%EBL), and rate of weight loss. Tertiary outcomes were to compare the incidence of symptomatic and asymptomatic gall bladder stone and timing in which gallstones symptomatize.in cases with laparoscopic sleeve gastrectomy with no concomitant laparoscopic cholecystectomy.

Method:

Preoperative work up included bariatric surgeons and nutritionists combining deliberation. Preoperative ultrasonography was performed in all patients. Preoperative anesthetist's appraisal. With induction of anesthesia, metronidazole 500 mg and ceftriaxone 1gm. given intravenously. Thrombotic prophylaxis with Clexane 4000 UI.

General anesthesia with the preservation of the air passage from soaking with heave. All measures were performed in mono-center in our unit for duration of 3 years by 3 surgeons competent in laparoscopic bariatric and biliary surgery ensuing the basics of bariatric and biliary surgeries. Each surgeon had preceding practice of at least 100 laparoscopic sleeve gastrectomies. At least one of three senior surgeons was always present to certify the same technique and inclusion criteria. Laparoscopic Sleeve Gastrectomy was performed in the classical steps [14].Following finalization of sleeve gastrectomy, the right upper quadrant was explored for the ongoing cholecystectomy. Cholecystectomy was accomplished using the same trocars and instruments used for the primary procedure. No added trocar was situated. Dissection of the gallbladder was performed using the ordinary monopolar diathermy. The gallbladder was delivered from the abdominal cavity through the 15-mm trocar incision. After completion of the procedure, tube drain was placed in the proximity of the gastric cut and another one in gall bladder bed.

On the second day after surgery, the patients could drink a little water. On the third day, upper gastrointestinal gastrograffin examinations were performed to rule out leakage. The peritoneal drainage tube was removed when the volume of peritoneal drainage was less than 15 mL. Patients were sanctioned to eat a semi-solid diet and were gradually proceed to a normal diet over the next 2-4 weeks.

All patients were followed for 1 month, 3 month, 6 month, 12 month and 24 months after hospital discharge. After discharge, patients were interacted with phone and follow up visit at outpatient clinic. Methods of follow up include full history and clinical examination to detect delayed drawbacks. At each office visit, body weight, body mass index (BMI), and gallstone-related symptoms were supervised. No patients lost during follow up period. Patients who missed the follow-up appointment in outpatient clinic were contacted via telephone and/or mail.

Statistical analysis:

The Collected data were statistically analyzed using Statistical Package for Social Science software (SPSS) (Version 20.0. Armonk, NY: IBM Corp). Continuous variables with a normal distribution were reported as mean and standard deviation (SD). Categorical variables were summarized as frequencies and percentages. Quantitative data with normal distribution was evaluated using Independent t-test between different groups and using Repeated Measures ANOVA with Paired t-test in the same group, while qualitative data was evaluated by Chi square test (χ2). Regression analysis was used to determine the independent factors affecting gallstone formation. Kaplan-Meier was used to analyze the survival rate of gallstone symptom-free. P values ≤0.05* and ≤0.001** were considered statistically significant and highly statistical significant respectively.

Discussion Coşkun etal, revealed concomitant cholecystectomy with laparoscopic sleeve gastrectomy lengthens the surgical span by 18-49 min .Other repelled concomitant cholecystectomy as this adds additional laparoscopy incisions .Moreover, Raziel et al, believed that concomitant cholecystectomy increased surgical span without an increase in days of stay after operation . Fuller etal, declared that concomitant cholecystectomy had devastating complications as high as 2%to 3%of cases . In our study, we agree that prolonged surgery is a drawback and we found to be nearly longer by 40.7min and increase postoperative hospital stay is another disadvantage however, we do not agree as regard additional incision. Although additional of 5 mm incisional is not a matter of importance but in our study we did not use any additional incision. The liver retractor in epigastrium was used to retract the liver and the two working instruments of laparoscopic sleeve were used to remove gall bladder. We found no statistically significant difference between both groups as regard intraoperative and postoperative complications in both groups. Mortality rate in group A was 2 % but no statistically significant difference. Also intraoperative and postoperative complications in concomitant cholecysteomy and cases with delayed cholecystectomy after sleeve are nearly the same with no advantages of one over the other so, no need to delay the laparoscopic cholecystomy and expose patients for another operation.

Raziel etal commented that concomitant cholecystectomy resulted in devastating complication as bile leakage . We found that bile leakage occurred in 2 cases only (2%) in group A and no statistically significant difference between both groups. Moreover, bile leakage occurred in 2 cases (3%) in cases of group B required surgery after sleeve gastrectomy. intraoperative and postoperative results are nearly the same whether cholecystectomy operated at the time of lap sleeve or deferred later on when gall stone symptomatizing required laparoscopic cholecystectomy.

The incidence of complicated gall bladder stones after laparoscopic sleeve gastrectomy varies between different studies. Sioka et al. validated to be 13.0% [17] and Festi et al. showed that the incidence may be 10% . On the contrarily, Li VK etal, declared that the incidence may reach up to 28% of patients However, in our study, the incidence of symptomatic gall bladder stone following sleeve gastrectomy is higher than stated by previous studies (55%) and 94 patients(85% of cases) occurred in the first year after sleeve and required another operation of laparoscopic cholecystectomy with big burden on patients. The high incidence of symptomatizing gall bladder stone after sleeve gastrectomy may be attributed to rapid weight loss within one year and regular follow up with close observation and ultrasonography that detect many cases with minimal symptoms. Our opinion is supported by other study .

In a study of 34 patients who developed symptomatic cholelithiasis within 2 years after bariatric surgery, 20 patients (58.2%) presented with acute cholecystitis. Laparoscopic cholecystectomy was changed to an open approach in 6 patients (17.6%) due to extensive adhesions or uncontrolled hemorrhage from the gallbladder bed . Furthermore, Amaral andThompson proposed a 27.6% incidence of complications related to gallstones after bariatric surgery, including common duct stones and pancreatitis. In our study, 26 cases (23%) presented with the commonest presentation of acute cholecystitis not improving on conservative treatment and required surgery within 72 hours. Laparoscopic cholecystectomy was converted to open cholecystectomy in 3 cases(5%) mostly due to bile leakage in 2 cases(3%) while tissue adhesion in one case(2%). conversion to open cholecystectomy in cases of concomitant cholecysteomy with sleeve occurred also in one case(1%) and in 3 cases (3%) due to biliary leakage. biliary leakage is the commonest cause of conversion due to familiarity of biliary system with anatomical aberration. however, we do not agree with the opinion in that adhesion post sleeve may increase morbidity of subsequent cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male and Non pregnant female, >20 years old, All patients were contender for bariatric surgery in conformity with National Institutes of Health consensus criteria for the management of morbid obesity (BMI ≥ 40 kg/m² or BMI ≥ 35 kg/m² with compelling co-morbidities linked to obesity),, had pre-operative ultrasound patients who completed at least two-years follow up

Exclusion Criteria:

* younger than 20 years, History of cholecystectomy, No pre-operative imaging available within 6 months, dearth of interest. Subjective mess and cognitive vulnerability that halt the patient from considering the operation, Drug or alcohol junkie, Patients unsuitable for general anesthesia, preceding bariatric operation, Patients with calcular obstructive jaundice underwent ERCP with stenting and Cases with arduous displaying of right upper quadrant or liver cirrhosis found at surgery.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
time of operation | 2 years
  time of operation in minutes
hospital length of stay | 2 years
  hospital length of stay i days

SECONDARY OUTCOMES:
body mass loss | 2 years
  percent excess body mass index loss

OTHER OUTCOMES:
timing in which gallstones symptomatize | 2 years
  timing in which gallstones symptomatize

IPD SHARING:
Plan to Share IPD: No